CLINICAL TRIAL: NCT01164150
Title: Prospective Randomised Phase II Trial Evaluating Adjuvant Pelvic Radiotherapy Using Either IMRT or 3-Dimensional Planning for Endometrial Cancer
Brief Title: Prospective Randomised Phase II Trial Evaluating Adjuvant Pelvic Radiotherapy Using Either IMRT or 3-Dimensional Planning for Endometrial Cancer. ICORG 09-06
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 09-06; CTRIAL-IE (ICORG) 09-06; EU-21048
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Endometrial Cancer; Gastrointestinal Complications; Radiation Toxicity; Urinary Complications
Keywords: gastrointestinal complications; urinary complications; radiation toxicity; recurrent endometrial carcinoma; endometrial adenocarcinoma; stage IA endometrial carcinoma; stage IB endometrial carcinoma; stage II endometrial carcinoma; stage IIIA endometrial carcinoma; stage IIIB endometrial carcinoma; stage IIIC endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Radiation Injuries

ARMS (2):
- Arm B (Experimental): Radiation: 45 Gy / 25 fractions pelvic radiotherapy using intensity modulated radiotherapy (IMRT) followed by 11 Gy / 2 fractions vaginal vault brachytherapy
  Interventions: Radiation: 45 Gy/25 fractions
- Arm A Control (Other): Radiation: 45 Gy/25 fraction external beam pelvic radiotherapy delivered using a 3-dimensional planned technique followed by 11 Gy / 2 fractions vaginal vault brachytherapy
  Interventions: Radiation: 45 Gy/25 fractions

INTERVENTIONS:
Radiation: 45 Gy/25 fractions — Arm A 45 Gy/25 fractions pelvic radiotherapy using 3D planned technique followed by 11Gy/2 fractions vaginal vault brachytherapy

SUMMARY:
Post-operative radiotherapy is internationally accepted as standard practice in the management of high-risk endometrial cancer1. Whilst it has no proven impact on overall survival it significantly increases local control.

Conventional radiotherapy techniques (3-dimensional) utilise a 3 or 4 field beam arrangement to target the pelvis in order to treat those areas at risk of recurrence: the vagina, the parametrium and the pelvic lymph nodes. However, when using such a technique it is not possible to avoid irradiating sensitive normal tissues such as the bowel and bladder.

Toxicity data from international randomised control trials in endometrial cancer report significantly more haematological, gastrointestinal, genitourinary and cutaneous toxicites (all grades) in those who received pelvic irradiation compared to those who did not2,3. These trials delivered radiotherapy using 2 or 3-dimensional techniques.

Intensity Modulated Radiation Therapy (IMRT) is a newer but established radiotherapy technique in many tumour sites that allows us to much more tightly conform the radiation. It uses computer-generated beams to produce radiotherapy volumes that can avoid irradiation of normal tissues in the pelvis.

There are no randomised studies reported in the literature that compare 3-dimensional pelvic irradiation with IMRT in patients who have had surgery for endometrial cancer. However there are several small studies that report considerable sparing of normal tissues using IMRT and when compared retrospectively with conventionally treated patients demonstrate marked reductions in acute gastrointestinal and genitourinary toxicity4.

By delivering post-operative radiotherapy to the pelvis using IMRT (as opposed to the standard 3-dimensional technique) it is anticipated that whilst local control and survival will be unaffected acute and late toxicity will be reduced.

DETAILED DESCRIPTION:
Primary Objective:

• To compare the incidence of acute grade >2 GU and GI toxicity

Secondary Objectives:

* To establish in the context of a clinical research study the feasibility of implementing pelvic nodal irradiation using IMRT in gynaecological cancer
* To establish an Image-Guided pathway for gynaecological cancer radiotherapy incorporating

  * Set-up errors and optimal margins for set-up uncertainty
  * Investigation of effects of bladder filling and rectal preparation protocols on the planning target volume
* To estimate the rate of loco-regional control
* To evaluate Quality of Life
* To estimate the rate of disease-free survival
* To estimate the overall survival rate
* To compare the incidence of late GU and GI toxicity

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing adjuvant pelvic radiotherapy for histologically confirmed endometrial adenocarcinoma / serous carcinoma / papillary serous carcinoma / mixed histology (adenocarcinoma and serous) and following AJCC 2009 grade/stage:

  * Grade 2: stage IB (LVSI +/or >60yrs)
  * Grade 3: stage IA and IB
  * Grade 1-3: Stage II and IIIA, IIIB and IIIC1
* Surgery consisting of total hysterectomy, +/- bilateral salpingo-oophorectomy, +/- lymph node sampling
* Staging with imaging of pelvis and abdomen (either MRI or CT)
* ECOG PS 0-2
* Age ≥ 18 years
* Provision of written informed consent in line with ICH-GCP guidelines

Exclusion Criteria:

* Previous radiotherapy to the pelvic region
* Patients in whom concurrent chemotherapy in planned
* Patients with macroscopic disease in situ
* History of inflammatory bowel disease
* Previous hip replacement
* Previous bowel surgery (excluding appendectomy)
* Patients with other syndromes/conditions associated with increased radiosensitivity
* The patient has or had other co-existing malignancies within the past 5 years other than non-melanoma skin cancer
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study or if it is felt by the research / medical team that the patient may not be able to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Reduction in the incidence of ≥ grade 2 acute genitourinary (GU) and gastrointestinal (GI) toxicity according to NCI CTCAE v.3.0 | 2015

SECONDARY OUTCOMES:
Incidence of late GI and GU toxicity according to NCI CTCAE v.3.0 | 2015
Feasibility of implementing pelvic nodal irradiation using intensity-modulated radiotherapy in gynecological cancer | 2015
Establishment of an image-guided pathway for gynecological cancer radiotherapy | 2015
Rate of loco-regional control as assessed by CT scan, MRI, and biopsy | 2015
Quality of life as assessed using EORTC QLQ-C30 and EORTC QLQ Cervical Cancer Specific Module CX 24 questionnaires | 2015
Rate of disease-free survival | 2015
Overall survival rate | 2015

CONTACTS AND LOCATIONS:
Overall Officials: Charles Gillham, Dr, Principal Investigator — Saint Luke's Hospital
Locations (5):
- Ireland (5):
  - St Luke's Radiation Oncology Network (SLRON) Centres, Dublin
  - St Luke's Centre for Radiation Oncology at Beaumont Hospital, Dublin
  - St Luke's Centre for Radiation Oncology at St James Hospital, Dublin
  - St Luke's Centre for Radiation Oncology at St Lukes Hospital, Dublin
  - Mid-Western Radiation Oncology Centre, Limerick